CLINICAL TRIAL: NCT00672048
Title: Expanding Quality Care for Glaucoma Through a Provider-Patient Partnership
Brief Title: Partnership for Glaucoma
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Duke University (Other)
Collaborators: University of Alabama at Birmingham (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: Pro00002593; R01EY018405-01 (NIH); NCT01733498 (obsolete NCT alias)
Record Dates: First submitted 2008-05-04; First posted 2008-05-06 (Estimated); Last update posted 2014-01-06 (Estimated); Status verified 2013-12

CONDITIONS: Glaucoma
Keywords: glaucoma; optometrists
MeSH Terms: conditions — Glaucoma

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Other)
  Interventions: Other: Computer Tablet; Other: Continuing Education Course
- 2 (Other): Control group to receive annual continuing education
  Interventions: Other: Continuing education

INTERVENTIONS:
Other: Computer Tablet — A tablet computer based software application designed to collect structured clinical information from providers and patients at the point of care.
  Arms: 1
Other: Continuing Education Course — Annual standard continuing education
  Arms: 1
Other: Continuing education — Annual standard continuing education materials
  Arms: 2

SUMMARY:
The purpose of this study is to develop new ways of assisting patients with glaucoma and their eye doctors in using the recommendations from practice guidelines.

DETAILED DESCRIPTION:
Glaucoma is a leading cause of blindness and visual impairment in the United States, particularly among disadvantaged populations. Despite the presence of therapies proven in NEI, randomized controlled trials that can be delivered by more than 18,000 ophthalmologists and 34,000 optometrists, almost nothing is known about the content and quality of glaucoma care delivered by non-MD providers such as optometrists. With the numbers of people with glaucoma expected to more than double in the next twenty years in the face of no more than a 15% increase in the supply of eye care providers, methods to better support appropriate and high-quality care for chronic eye diseases such as glaucoma delivered by optometrists will become as critical, if not more so, as techniques to enhance quality care among ophthalmologists.

Our study is a community-based, randomized, controlled trial that evaluates the suitability and effectiveness of a technology-based (tablet computer) intervention within the context of a novel partnership between optometrists and patients with glaucoma to improve the process quality of care and ultimately outcomes of care. By using successfully implemented technology in novel applications,and by building on the success of ongoing community-based quality improvement projects in our region, the study provides a means for rapid translation into community care if the intervention is successful.

ELIGIBILITY:
Inclusion Criteria:

-Diagnosis of open angle glaucoma with documented visual field loss.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 721 (Actual)
Dates: Start 2007-10; Primary Completion 2013-07 (Actual); Study Completion 2013-07 (Actual)

PRIMARY OUTCOMES:
To determine if innovative technology will improve process quality of care & important outcomes of care by optometrists in a cost-efficient manner while simultaneously empowering & including patients as part of the care process. | Baseline, Year 1 and Year 2

CONTACTS AND LOCATIONS:
Overall Officials: Paul Lee, MD, JD, Principal Investigator — Duke University
Locations (2):
- United States (2):
  - University of Alabama, Birmingham, Alabama
  - Duke University, Durham, North Carolina

REFERENCES:
- [Background] Silvey GM, Lobach DF, Macri JM, Hunt M, Kacmaz RO, Lee PP. User interface considerations for collecting data at the point of care in the tablet PC computing environment. AMIA Annu Symp Proc. 2006;2006:1096. PMID 17238715
- [Background] Silvey GM, Lobach DF, Macri JM, Hunt M, Kacmaz RO, Lee PP. Overcoming obstacles to collecting narrative data from eye care professionals at the point-of-care. AMIA Annu Symp Proc. 2005;2005:1116. PMID 16779403
- [Background] Kacmaz RO, Arbanas JM, Lee PP, Lobach DF. Assessment of relative importance of tablet computer features in supporting direct electronic documentation of encounters by eye care professionals. AMIA Annu Symp Proc. 2005;2005:1001. PMID 16779288
- [Background] Lobach DF, Silvey GM, Macri JM, Hunt M, Kacmaz RO, Lee PP. Identifying and overcoming obstacles to point-of-care data collection for eye care professionals. AMIA Annu Symp Proc. 2005;2005:465-9. PMID 16779083